CLINICAL TRIAL: NCT04187001
Title: Home Exercises for Neck Pain: a Delphi Survey
Brief Title: Home Exercises Protocol for Neck Pain
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Laylla Marjorye Rebouças Bezerra, Laylla Marjorye, Universidade Federal de Pernambuco
Other Study IDs: 3.007.662
Record Dates: First submitted 2019-12-02; First posted 2019-12-05 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Neck Pain
Keywords: stabilization; exercise; Delphi
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Judges: Professionals that assess the content validity of the exercise protocol
  Interventions: Other: Content Validity
- Target population: People that assess the exercise protocol for cultural adaptation
  Interventions: Other: Cultural adaptation

INTERVENTIONS:
Other: Content Validity — Use Delphi technique for achieve consensus
  Groups: Judges
Other: Cultural adaptation — Adapt the content to the target population
  Groups: Target population

SUMMARY:
Delphi study about home exercise protocol development for neck pain.

DETAILED DESCRIPTION:
Introduction: Neck pain is rising globally as a musculoskeletal disorder, as a result of several factors. Currently, there are several types of treatments for cervicalgia, applied according to the therapist's choice and patient's conditions and preferences, however, there are no reports of an effective self-performing treatment aiming to stabilizing the cervical, giving musculoskeletal balance, and focus on reducing pain.

It is important the promotion of a self-performing treatment, resulting in a high cost benefit because patient does not have to move to perform the treatment outside his or her home, does not need financial resources and demands little time to perform it. In addition to decreasing the frequency and intensity of hospitalizations and government costs incurred in this musculoskeletal disorder. Therefore, the study aims to construct, validate and adapt a self-performing exercise protocol in reducing cervical pain.

Methods: The first phase was the development of the first version of the protocol, through literature search; in the second phase, the content was validated, through evaluation by a committee of nine physiotherapists judges using the Delphi technique; and the last phase of the protocol, the cultural adequacy, is being performed through evaluation by fifteen participants of the target population to assemble the final version of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Judges: physical therapists with at least 2 years of experience in cervical area.
* Target population: chronic neck pain.

Exclusion Criteria:

* Vestibular system problems, balance impairment, nervous system-related disorders, inability to perform exercises, history of cervical trauma or surgery in the region, history of cervical radiculopathy, history of cervical spine injury, temporomandibular dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physical therapists with publication or experience in cervical area. Individuals with chronic neck pain.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-05-13 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Concordance | february - may 2019
  degree of consensus by percentage, content validity index

CONTACTS AND LOCATIONS:
Overall Officials: Gisela R Siqueira, PhD, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bezerra LMR, Melo TMS, Gomes VMDSA, Pas RCD, Alves LIDN, Salemi MM, Silva IR, Tenorio ADS, Siqueira GR. Home exercises for neck pain: A Delphi survey. Physiother Res Int. 2023 Apr;28(2):e1982. doi: 10.1002/pri.1982. Epub 2022 Nov 14. PMID 36373555